CLINICAL TRIAL: NCT00478829
Title: Prevalence of Depression and Anxiety in Patients Seeking Medical Care at General Health Care Settings in 5 Large Cities in China
Brief Title: Prevalence of Depression and Anxiety in Patients Seeking Medical Care at General Health Care Settings in China
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 0600B2-4417
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Adult

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Objectives: Primary: To estimate the prevalence of depression and/or anxiety disorder in outpatients attending the general health care settings in China.

Secondary:

* To estimate gender- and age-specific prevalence of depression and/or anxiety disorder in outpatients attending the general health care settings in China.
* To estimate the prevalence of depression and/or anxiety disorder in outpatients attending the general health care settings such as departments of neurology, gastroenterology, cardiology, and gynecology.
* To describe the recognition and treatment rate by treating physicians as depression and/or anxiety for outpatients in the general health care settings in China.

DETAILED DESCRIPTION:
This study is designed to investigate the status of identifying depression and/or anxiety disorder with somatic symptoms in general hospitals in China. The study will generate valuable information to the medical community; therefore the early and vigorous treatment is possible. It's in line with China government authorities' target to increase the recognition rate of depression and/or anxiety in primary care settings to more than 50% by the end of 2010. The study will also help to identify specific diagnosis and treatment patterns for depressive / anxious patients and their comorbid conditions.

ELIGIBILITY:
Main Inclusion Criteria:

* Greater than or equal to 18 years.
* Consecutive general internal medical outpatients attending the selected general hospitals in the investigate days(Department of neurology, gastrointestinal, cardiology and gynecology).
* Informed consent obtained for all patients who will undergo a standardized diagnostic assessment by specialized psychiatrists.

Main Exclusion Criteria:

* Patients who have been screened on a previous visit.
* Patients who are unable to complete the survey because of mental or physical incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000
Dates: Start 2007-04; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For China, medinfo@wyeth.com
Locations (5):
- China (5):
  - Beijing, Beijing Municipality
  - Guangzhou, Guangdong
  - Changsha, Hunan
  - Shanghai, Shanghai Municipality
  - Chengdu, Sichuan